CLINICAL TRIAL: NCT02236312
Title: A Multicentre, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Three Doses of Botulinum Toxin in the Treatment of Moderate to Very Severe Glabellar Frown Lines
Brief Title: Safety and Efficacy Study of Botulinum Toxin for the Treatment of Glabellar Frown Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43QM1313
Record Dates: First submitted 2014-09-01; First posted 2014-09-10 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2016-05

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Botulinum Toxin 30 units (Experimental): I.M. injection
  Interventions: Drug: Botulinum Toxin Type A
- Botulinum Toxin 45 units (Experimental): I.M. injection
  Interventions: Drug: Botulinum Toxin Type A
- Botulinum Toxin 60 units (Experimental): I.M. injection
  Interventions: Drug: Botulinum Toxin Type A
- Placebo (Placebo Comparator): I.M. injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A
  Arms: Botulinum Toxin 30 units; Botulinum Toxin 45 units; Botulinum Toxin 60 units
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy in wrinkle reduction of a single treatment of three different doses of botulinum toxin compared to placebo, in the treatment of moderate to very severe glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to Very Severe glabellar lines at maximum frown as assessed by the subject and the Investigator and at least Mild glabellar lines at rest

Exclusion Criteria:

* Any previous treatment with any botulinum toxin
* Rhytids of the glabellar region that cannot be smoothed out by manually spreading the skin apart
* Any previous insertion of any permanent or semi-permanent material, hyaluronic acid or collagen fillers to the glabellar region
* Any history of facial surgery above the lower orbital rim
* Any planned facial surgery or aesthetic procedure during the study period
* Ablative skin resurfacing or chemical peels above the lower orbital rim in the previous 12 months or during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Reduction of glabellar frown line severity on Day 14 following treatment with botulinum toxin | 14 Days
  Reduction in glabellar frown line severity is derived separately for the Investigator and the subject assessment, using a validated photo scale, at maximum frown on Day 14.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Private practice, Birmingham, Alabama
  - Private practice, Mobile, Alabama
  - Private practice, San Diego, California
  - Private practice, Englewood, Colorado
  - Private practice, Aventura, Florida
  - Private practice, Nashville, Tennessee
  - Private practice, San Antonio, Texas
  - Private practice, Salt Lake City, Utah